CLINICAL TRIAL: NCT06554821
Title: An Open-label, Randomised, Parallel-group, Fixed-sequence Study to Assess the Effect of Oral Ticagrelor on the Pharmacokinetics of Oral Rosuvastatin in Healthy Participants
Brief Title: A Study to Investigate the Effect of Oral Ticagrelor on the Pharmacokinetics of Oral Rosuvastatin When Given in Healthy Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Collaborators: Parexel (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: D3560C00817
Record Dates: First submitted 2024-08-02; First posted 2024-08-15 (Actual); Last update posted 2025-04-18 (Actual); Status verified 2025-04

CONDITIONS: Healthy Participants
Keywords: Rosuvastatin; Ticagrelor; Pharmacokinetics
MeSH Terms: interventions — Rosuvastatin Calcium; Ticagrelor

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Rosuvastatin (Dose 1) + Ticagrelor (Experimental): Participants will receive rosuvastatin (dose 1) orally as a single dose on Day 1 in Period 1 and Day 6 in Period 2. During Period 2, participants will also receive ticagrelor 90 mg BID (twice a day) on Day 6 through Day 10.
  Interventions: Drug: Rosuvastatin; Drug: Ticagrelor
- Rosuvastatin (Dose 2) + Ticagrelor (Experimental): Participants will receive rosuvastatin (dose 2) orally as a single dose on Day 1 in Period 1 and Day 6 in Period 2. During Period 2, participants will also receive ticagrelor 90 mg BID on Day 6 through Day 10.
  Interventions: Drug: Rosuvastatin; Drug: Ticagrelor

INTERVENTIONS:
Drug: Rosuvastatin — Participants will receive rosuvastatin (dose 1 or dose 2) orally as a single dose on Day 1 in Period 1 and Day 6 in Period 2.
  Other Names: CRESTOR
Drug: Ticagrelor — Participants in each arm will receive ticagrelor 90 mg orally BID from Day 6 to Day 10.
  Other Names: BRILIQUE

SUMMARY:
The purpose of this study is to measure the effect of ticagrelor on the pharmacokinetics (PK) of rosuvastatin in healthy participants.

DETAILED DESCRIPTION:
This study will be conducted at a single Clinical Unit. It includes 2 parallel arms (one for each rosuvastatin dose) and 2 treatment periods.

The study will comprise:

* A Screening Period of maximum 28 days.
* Period 1: It will start on Day -1. A single dose of rosuvastatin (dose 1 or dose 2) will be administered on Day 1 followed by PK sampling of rosuvastatin for 96 hours. Participants will be admitted to the Clinical Unit on Study Day -1. Period 1 will end on Study Day 5.
* Period 2: It will start on Study Day 6. A second single dose of rosuvastatin (dose 1 or dose 2) will be administered on Day 6 followed by PK sampling of rosuvastatin for 120 hours. Ticagrelor 90 mg, twice a day will be started on Day 6 (administered concomitantly with rosuvastatin) and administered through Day 10. Period 2 will end on Study Day 12.
* A Follow-up Visit, 4 to 7 days after discharge.

ELIGIBILITY:
Inclusion Criteria:

* Healthy participants with suitable veins for cannulation or repeated venipuncture.
* All females must have a negative pregnancy test at the Screening Visit and on admission to the Clinical Unit.
* Females of childbearing potential must not be lactating and if heterosexually active must agree to use an approved method of highly effective contraception, to avoid pregnancy from the time of first administration of study intervention until 1 month after the study Follow-up Visit.
* Females of non-childbearing potential must be confirmed at the Screening Visit by fulfilling one of the following criteria:

  1. Postmenopausal defined as amenorrhea for at least 12 months following cessation of all exogenous hormonal treatments and follicle-stimulating hormone (FSH) levels in the postmenopausal range.
  2. Documentation of irreversible surgical sterilization by hysterectomy, bilateral oophorectomy, or bilateral salpingectomy but not tubal ligation or tubal occlusion.
* Sexually active fertile male participants with partners of childbearing potential must adhere to the specified contraception methods from the time of first administration of study intervention administration until 2 weeks after the study Follow-up Visit.
* Have a BMI between 18 and 30 kg/m2 inclusive and weigh at least 50 kg and no more than 100 kg inclusive.

Exclusion Criteria:

* History of any clinically important disease or disorder which may either put the participant at risk or influence the results or the participant's ability to participate in the study.
* History or presence of gastrointestinal, hepatic, or renal disease or any other condition known to interfere with absorption, distribution, metabolism, or excretion of drugs.
* Any clinically important illness, medical/surgical procedure, or trauma within 4 weeks of the first administration of study intervention.
* Any clinically important abnormal laboratory values or vital signs.
* Any positive result on Screening for serum HBsAg OR anti-HBc antibody, indicative of active hepatitis B (i.e., participants with positive anti HBc antibody result are acceptable if anti HBc IgM antibodies are negative).
* Current smokers or those who have smoked or used nicotine products (including e-cigarettes) within the previous 3 months prior to screening.
* Known or suspected history of alcohol or drug abuse or excessive intake of alcohol. Excessive intake of alcohol defined as the regular consumption of more than 24 g of alcohol per day for men or 12 g of alcohol per day for females.
* Positive screen for drugs of abuse, or alcohol or cotinine at screening or on admission to the Clinical Unit.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 28 (Actual)
Dates: Start 2024-08-05 (Actual); Primary Completion 2024-10-08 (Actual); Study Completion 2024-10-08 (Actual)

PRIMARY OUTCOMES:
Area under concentration-time curve from time 0 to infinity (AUCinf) | From Day 1 to Day 11
  To assess the effect of ticagrelor on plasma PK (AUCinf) of rosuvastatin dose 1 and dose 2 separately, in healthy participants.
Area under concentration-curve from time 0 to the last quantifiable concentration (AUClast) | From Day 1 to Day 11
  To assess the effect of ticagrelor on plasma PK (AUClast) of rosuvastatin dose 1 and dose 2 separately, in healthy participants.
Maximum observed drug concentration (Cmax) | From Day 1 to Day 11
  To assess the effect of ticagrelor on plasma PK (Cmax) of rosuvastatin dose 1 and dose 2 separately, in healthy participants.

SECONDARY OUTCOMES:
Number of participants with adverse events (AEs) | Approximately 7 weeks
  To examine the safety and tolerability of rosuvastatin alone and in combination with ticagrelor.
Terminal elimination half-life (t1/2) | From Day 1 to Day 11
  To assess the effect of ticagrelor on the PK (t1/2) of rosuvastatin in healthy participants.
Terminal rate constant (parent only) (λz) | From Day 1 to Day 11
  To assess the effect of ticagrelor on the PK (λz) of rosuvastatin in healthy participants.
Time to reach maximum observed concentration (tmax) | From Day 1 to Day 11
  To assess the effect of ticagrelor on the PK (tmax) of rosuvastatin in healthy participants.
Amount of drug excreted (Ae) | From Day 1 to Day 11
  To assess the effect of ticagrelor on the urine PK (Ae) of rosuvastatin in healthy participants.
Renal clearance (Clrenal) | From Day 1 to Day 11
  To assess the effect of ticagrelor on the urine PK (Clrenal) of rosuvastatin in healthy participants.
Percent of dose excreted | From Day 1 to Day 11
  To assess the effect of ticagrelor on the urine PK of rosuvastatin in healthy participants.

CONTACTS AND LOCATIONS:
Locations (1):
- Research Site, Berlin, Germany

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymized individual patient-level data from AstraZeneca group of companies sponsored clinical trials via the request portal Vivli.org. All requests will be evaluated as per the AZ disclosure commitment: https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
  "Yes", indicates that AZ are accepting requests for IPD, but this does not mean all requests will be approved.
Time Frame: AstraZeneca will meet or exceed data availability as per the commitments made to the EFPIA/PhRMA Data-Sharing Principles. For details of our timelines, please refer to our disclosure commitment at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
Access Criteria: When a request has been approved AstraZeneca will provide access to the anonymized individual patient-level data via secure research environment Vivli.org. A Signed Data Usage Agreement (non-negotiable contract for data accessors) must be in place before accessing requested information.
URL: https://vivli.org/